CLINICAL TRIAL: NCT05648032
Title: The Clinical Application of PLT Combined With Steroid in Lateral Epicondylopathy and Supraspinatus Calcific Tendinopathy
Brief Title: PLT and Steroid in Lateral Epicondylopathy and Supraspinatus Calcific Tendinopathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201903076DIPC
Record Dates: First submitted 2022-11-20; First posted 2022-12-13 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-04

CONDITIONS: Lateral Epicondylitis; Rotator Cuff Syndrome
MeSH Terms: conditions — Tennis Elbow | interventions — Triamcinolone Acetonide; Steroids

STUDY DESIGN:
Intervention Model Description: Tennis elbow Supraspinatus calcific tendinitis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The syringe is covered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLT (lyophilized platelet) with steroid (Experimental): PLT (30ng)+1.0 mL 1.0% Lidocaine+1.0 mL (10.0 mg/mL) Triamcinolone acetonide, once
  Interventions: Combination Product: lyophilized platelet (30ng) and triamcinolone acetonide 10mg
- PLT (lyophilized platelet) (Experimental): PLT (30ng)+1.0 mL 1.0% Lidocaine+1.0 mL normal saline, once
  Interventions: Other: lyophilized platelet (30ng)
- Steroid (Active Comparator): 1.0 mL 1.0% Lidocaine+1.0 mL (10.0 mg/mL) Triamcinolone acetonide, once
  Interventions: Drug: triamcinolone acetonide 10mg

INTERVENTIONS:
Combination Product: lyophilized platelet (30ng) and triamcinolone acetonide 10mg — Ultrasound-guided injection of lyophilized platelet (30ng)+1.0 mL 1.0% Lidocaine+1.0 mL (10.0 mg/mL) Triamcinolone acetonide into the hypoechoic area of common extensor tendon (in lateral epicondylopathy) or around calcific spots (in supraspinatus calcific tendinitis)
  Other Names: PLT and steroid
  Arms: PLT (lyophilized platelet) with steroid
Other: lyophilized platelet (30ng) — Ultrasound-guided injection of PLT (30ng)+1.0 mL 1.0% Lidocaine+1.0 mL normal saline into the hypoechoic area of common extensor tendon (in lateral epicondylopathy) or around calcific spots (in supraspinatus calcific tendinitis)
  Other Names: Blood product
  Arms: PLT (lyophilized platelet)
Drug: triamcinolone acetonide 10mg — Ultrasound-guided injection of 1.0 mL 1.0% Lidocaine+1.0 mL (10.0 mg/mL) Triamcinolone acetonide into the hypoechoic area of common extensor tendon (in lateral epicondylopathy) or around calcific spots (in supraspinatus calcific tendinitis)
  Other Names: steroid
  Arms: Steroid

SUMMARY:
PLT vs. steroid vs. PLT + steroid, which treatment is most effective in lateral epicondylitis (or tennis elbow) and supraspinatus calcific tendinitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (or tennis elbow) and supraspinatus calcific tendinitis are common tendinopathies of the upper limb and both have negative impacts on the patients' quality of life. The former affects function of wrist extension due to degeneration of common extensor tendons; the latter causes severe pain and limitation of shoulder range of motion due to calcific deposits within the supraspinatus tendon. Current common injection therapies are ultrasound-guided injection of steroid or platelet-rich plasma (PRP).

Previous studies have shown that steroid injection provides early but short-term pain reduction, while PRP injection causes post-injection pain by inducing inflammation but provides long-term pain relief and functional improvement. It may provide early pain reduction with long-term tissue regeneration if combining steroid and PRP. A recent study on tennis elbow showed that inclusion of steroid in the autologous whole blood and 20% dextrose injection can reduce pain during early treatment, without interfering with the therapeutic effects.

Furthermore, disadvantages of current PRP include difficulty in quantifying platelet numbers and growth factor activity, and in long-term preservation. In this study lyophilized platelet (PLT) can solve these problems, which can be dissolved in saline before injection.

This 3-arm randomized controlled trial will divide subjects into the PLT group (group A), steroid group (group B) or PLT+steroid group (group C). Therapeutic effects will be evaluated by pain visual analogue scale (VAS), grip dynamometer, and disabilities of the arm, shoulder, and hand (DASH) questionnaires during follow-ups at 2nd, 4th, 6th, 12th and 24th week after treatment, and ultrasound at 12th and 24th week . The hypothesis is that PLT+steroid injection will have earlier pain reduction than PLT injection and longer effects of pain reduction and functional improvement.

ELIGIBILITY:
Lateral epicondylitis

Inclusion Criteria:

* Tenderness at lateral epicondyle more than 3 months
* Ultrasound-confirmed lateral epicondylopathy
* Pain VAS ≥ 3/10 during wrist resistive extension
* No treatment response to NSAID and physiotherapy

Exclusion Criteria:

* Pregnancy or lactation
* Carpal tunnel syndrome (the same arm) in one year
* Cervical radiculopathy
* Taking NSAID in one week
* Receiving PRP or steroid injection in one month
* History of bacteremia, cellulitis or skin ulcer in three months
* Rheumatoid arthritis
* Malignancy
* Poorly controlled diabetets mellitus (DM), liver and kidner diseases
* Severe anemia (Hb<5)
* Thrombocytopenia
* History of tennis elbow surgery
* History of elbow trauma

Supraspinatus calcific tendinis

Inclusion Criteria:

* Hawkins-Kennedy test or empty can test, one of which is positive
* Ultrasound-confirmed (calcification > 2mm)
* Pain VAS ≥ 3/10 over right deltoid area more than 3 months
* No treatment response to NSAID and physiotherapy

Exclusion Criteria:

* Pregnancy or lactation
* Carpal tunnel syndrome (the same arm) in one year
* Cervical radiculopathy
* Taking NSAID in one week
* Receiving PRP or steroid injection in one month
* History of bacteremia, cellulitis or skin ulcer in three months
* Rheumatoid arthritis
* Malignancy
* Poorly controlled DM, liver and kidner diseases
* Severe anemia (Hb<5)
* Thrombocytopenia
* History of shoulder surgery
* History of shoulder trauma

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Lateral elbow pain and shoulder pain (worst in the last one week) | 24 weeks post-injection
  Visual analogue scale (0-10, the high the worse)

SECONDARY OUTCOMES:
Lateral elbow pain and shoulder pain (worst in the last one week) | Baseline, 2, 4, 6, and 12 weeks post-injection
  Visual analogue scale (0-10, the high the worse)
Functional | Baseline, 2, 4, 6, 12, and 24 weeks post-injection
  Disabilities of the Arm, Shoulder, and Hand (Score 0-100, the high the worse)
Grasping power | Baseline, 2, 4, 6, 12, and 24 weeks post-injection
  Grasping power
Ultrasound | Baseline, 12 and 24 weeks post-injection
  Tendon thickness (mm)
Ultrasound | Baseline, 12 and 24 weeks post-injection
  Calcification size (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Hung Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan